CLINICAL TRIAL: NCT05180214
Title: The Effect of Adding Ketorolac to Bupivacaine in Superficial Cervical Plexus Block in Thyroid Surgery.
Brief Title: Analgesia for Thyroidectomy Using Bilateral Superficial Cervical Plexus Block With Bupivacaine Only or Adding Ketorolac to it.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fouad Soliman, Lectuerer of Anesthesia and ICU, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2006
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Thyroid Goiter; Thyroid Nodule
Keywords: ketorolac, superficial cervical plexus block, thyroidectomy
MeSH Terms: conditions — Goiter; Thyroid Nodule | interventions — Bupivacaine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine (Active Comparator)
  Interventions: Drug: Bupivacain
- bupivacaine and ketorolac (Active Comparator)
  Interventions: Drug: Bupivacain; Drug: Ketorolac

INTERVENTIONS:
Drug: Bupivacain — analgesic
Drug: Ketorolac — analgesia
  Arms: bupivacaine and ketorolac

SUMMARY:
Thyroidectomy is considered a common operation with moderate to severe postoperative pain in some patients. Patients are divided into two groups. Bupivacaine group received bilateral superficial cervical plexus block (BSCPB) with 10 ml of bupivacaine (0.25%) and 1 ml of normal saline on each side and the Bupivacaine Ketorolac group received (BSCPB) with 10 ml of bupivacaine (0.25%) and 1 ml of ketorolac (15 mg) on each side.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-50 years
* ASA I-II patients
* Patients going to do thyroid surgeries under general anesthesia

Exclusion Criteria:

* Patient refusal
* Known history of sensitivity to the drug used in the study
* Drug abuse
* Infection at the site of the block
* Presence of coagulopathy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
1st analgesic requirement | 24 hours
  The first time of supplemental analgesic need postoperatively

SECONDARY OUTCOMES:
analgesic consumption | 24 hours
  total analgesic consumption
postoperative pain | 24 hours
  visual analogue scale(0-10) 0=no pain and 10=severe intolerable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Faculty of Medicine, Sohag, Egypt